CLINICAL TRIAL: NCT03121534
Title: A Phase II Study of Ibrutinib, Nivolumab and Blinatumomab in Richter Transformation
Brief Title: Ibrutinib, Nivolumab and Blinatumomab in Richter Transformation
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The study was closed for slow accrual
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2016-0765
Record Dates: First submitted 2017-04-14; First posted 2017-04-20 (Actual); Results first posted 2023-02-17 (Actual); Last update posted 2023-02-17 (Actual); Status verified 2023-01

CONDITIONS: Hematopoietic/Lymphoid Cancer; Richter's Transformation
Keywords: Hematopoietic/Lymphoid Cancer; Richter's transformation; RT; Blinatumomab; Dexamethasone; Decadron
MeSH Terms: conditions — Hematologic Neoplasms | interventions — blinatumomab; Dexamethasone; Calcium Dobesilate; ibrutinib; Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Ibrutinib, Nivolumab and Blinatumomab (Experimental): 2 (8week) cycles of ibrutinib, nivolumab and blinatumomab. 9 (4week) cycles ibrutinib and nivolumab. Maintenance with ibrutinib monotherapy until disease progression following completion of nivolumab.
  Ibrutinib treatment will begin cycle 1, day 1 at 420mg/d. Nivolumab for up to a total of 52 weeks. Dosing will be 240mg IV every 2 weeks, commencing on day 1 until 2nd response assessment, then 480mg IV every 4 weeks.
  blinatumomab continuous IV infusion, starting day 15 of cycle 1 and day 1 of cycle 2, for 2 courses of 4 weeks each separated by a 2 week blinatumomab treatment-free interval. Hospitalization in cycle 1 on day 15-31 (first 17 days of blinatumomab therapy). Blinatumomab will be initiated at 9mcg/day from day 15-21, followed by 28 mcg/day from day 22-28, followed by 112 mcg/day from day 29-42. In cycle 2, patients will be admitted for the first 3 days. Blinatumomab in cycle 2 will be administered at a dose of 112 mcg/day from day 1-28.
  Interventions: Drug: Blinatumomab; Drug: Dexamethasone; Drug: Ibrutinib; Drug: Nivolumab

INTERVENTIONS:
Drug: Blinatumomab — Patients will receive blinatumomab as a continuous IV infusion, commencing on day 15 of cycle 1 and day 1 of cycle 2, for 2 courses of 4 weeks each separated by a 2 week .
  blinatumomab will be initiated at 9mcg/day from day 15-21, followed by 28 mcg/day from day 22-28. This will be followed by 112 mcg/day from day 29-42. In cycle 2, patients will be admitted for the first 3 days.blinatumomab treatment-free interval.
  Other Names: BLINCYTO®
Drug: Dexamethasone — Dexamethasone 20 mg by mouth or vein 24 hours prior to and within 1 hour before start of treatment in each treatment cycle. If treatment is interrupted for >4 hours at any point, Dexamethasone treatment given before re-initiation of therapy. Dexamethasone 8 mg by mouth or vein every 8 hours given for 48 hours at the commencement of the infusion and after each dose increment.
  Other Names: Decadron
Drug: Ibrutinib — Ibrutinib treatment will commence on cycle 1, day 1 at 420mg/d. Dose reductions to 280mg/d or 140mg/d are allowed per treating physician discretion, but the reason must be documented in the medical record. Ibrutinib will be given continuously until disease progression or toxicity.
  Other Names: Imbruvica™
Drug: Nivolumab — Patients will receive nivolumab for up to a total of 52 weeks. Dosing will be 240mg IV every 2 weeks, commencing on day 1 until 2nd response assessment, then 480mg IV every 4 weeks.
  Other Names: Opdivo

SUMMARY:
The goal of this clinical research study is to learn if blinatumomab can help to control Richter Transformation (RT, a type of blood cancer). The safety of this drug will also be studied.

This is an investigational study. Blinatumomab is FDA approved and commercially available for the treatment of acute lymphoblastic leukemia (ALL). It is investigational to use blinatumomab to treat patients with RT. The study doctor can explain how the study drug is designed to work.

Up to 21 participants will be enrolled in this study. All will take part at MD Anderson.

DETAILED DESCRIPTION:
Study Drug Administration:

The study has 2 study cycles. Cycle 1 is 8 weeks, followed by a 4-8 week break, and then Cycle 2 is 4 weeks.

If you are found to be eligible to take part in this study, you will receive blinatumomab by a central venous catheter (CVC) continuously (non-stop) for 1-2 cycles, depending on how you are responding to the study drug. A CVC is a sterile flexible tube that will be placed into a large vein while you are under local anesthesia. Your doctor will explain this to you in more detail, and you will be required to sign a separate consent form for this procedure.

During Cycle 1, the blinatumomab infusion will be started in the hospital. You will be in the hospital for up to at least 16 nights/17 days so that you can be checked for side effects. During Cycle 2, the blinatumomab infusion will also be started in the hospital. You will be in the hospital for at least 2 nights/3 days. Your doctor will decide when you can leave the hospital. Also, if treatment is interrupted for more than 4 hours, for any reason, you will need to be admitted to the hospital to restart the treatment.

Blinatumomab will be delivered by a small pump, which you will carry with you for the whole time you receive the drug. You will be given a shoulder or belt bag to hold the pump and infusion bag. You will be able to wear regular clothes, walk around, and perform daily living activities. You will be given instructions for taking a shower and other activities. There will be some things that you should not do, such as go swimming. The study staff will give you more information on activities you should not do while receiving the drug.

You will need to come to MD Anderson to have the infusion bags changed every 48 hours. The study staff will let you know when you need to return to the clinic.

You will be given standard drugs, such as dexamethasone, to help decrease the risk of side effects. You may ask the study staff for information about how the drugs are given and their risks.

If you have severe side effects, your study doctor may decide to stop treatment permanently or temporarily. If you recover or if the symptoms have improved, the treatment may be continued. If the doctor thinks it is needed, you will have an MRI and possibly also a spinal tap (lumbar puncture) to test the fluid around the brain, before you restart treatment.

Length of Study:

You may receive blinatumomab for up to 2 cycles. You will no longer be able to take the study drug if the disease gets worse, if serious side effects occur, or if you are unable to follow study directions. Additionally, if your doctor feels it is in your best interests to receive an alternative treatment for your Richter Transformation, such as allogeneic stem cell transplantation, you will no longer be able to receive blinatumomab.

Your participation on this study will be over after you have completed follow-up.

Study Visits:

At any time the doctor thinks it is needed, you may have a neurological exam.

Based on the results of the below tests after Cycle 1, the study doctor will decide if you will continue to receive the study drug during Cycle 2. If you do not receive the drug during Cycle 2, you will have an end-of-study visit (described below).

On Days 1-17 of Cycle 1 (the time you are in the hospital), every week during Cycle 1, Days 1-3 of Cycle 2, and every week of Cycle 2:

* You will have a physical exam.
* Blood (about 2-3 teaspoons) will be drawn for routine tests.

About 2-4 weeks after Cycles 1 and 2:

* You will have a physical exam.
* Blood (about 2-3 teaspoons) will be drawn for routine tests.
* You will have a bone marrow biopsy/aspiration to check the status of the disease.
* You will have a PET/CT or CT scan.

About 24 weeks after the first dose of study drug and then every 12 weeks after that for up to 96 weeks:

* You will have a physical exam.
* Blood (about 2-3 teaspoons) will be drawn for routine tests.
* You will have a PET/CT or CT scan to check the status of the disease.

End-of-Study Visit:

After the last dose of study drug, you will continue to receive routine medical care as part of your standard care. However, if the disease comes back or worsens while you are receiving the study drug:

* You will have a physical exam.
* Blood (about 2-3 teaspoons) will be drawn for routine tests.
* You will have a bone marrow biopsy/aspiration
* You will have a PET/CT scan to check the status of the disease.
* If the doctor thinks it is needed, you may have a lymph node biopsy to confirm that the disease has come back.
* If you can become pregnant, blood (about 1 teaspoon) or urine will be collected for a pregnancy test.

Long-Term Follow-up:

After you have completed your participation in this study, you will be asked to participate in a separate leukemia department protocol (DR09-0223). The purpose of this protocol is to determine how long patients live after receiving leukemia treatment. On this study, if you are not having follow-up at MD Anderson, study staff will contact you via phone, email, or MyMDAnderson every 6-12 months, to see how you are doing. Phone calls will take approximately 5-10 minutes. If you agree, you will sign a separate consent form for this study.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with previously treated CLL and biopsy-proven Richter's transformation with DLBCL histology according to IWCLL criteria (Richter Transformation - RT) and CD19 positive by flow cytometry OR immunohistochemistry.
2. Eastern Co-operative Oncology Group (ECOG) performance status < or =2.
3. Age > or =18 years at the time of informed consent.
4. Able to provide informed consent and be willing to participate in study schedule and events.

Exclusion Criteria:

1. Other active malignancy receiving systemic therapy.
2. History or presence of clinically relevant disorder affecting the CNS such as epilepsy, childhood or adult seizure, paresis, aphasia, stroke, severe brain injuries, dementia, Parkinson's disease, cerebellar disease, organic brain syndrome, or psychosis, with the exception of a history of CNS lymphoma that is controlled with intrathecal therapy.
3. Known active DLBCL in the CNS (confirmed by CSF analysis).
4. Current autoimmune disease requiring >/= 20mg/day of prednisone or systemic immunosuppressive therapy (eg. with cyclosporine or azathioprine).
5. Allogeneic HSCT within 24 weeks before the start of protocol-specified therapy.
6. Active Graft-versus-Host Disease (GvHD), grade 2-4 according to the Glucksberg criteria, active chronic GvHD requiring systemic treatment or requirement for GvHD prophylaxis with cyclosporine or tacrolimus.
7. Cancer chemotherapy within 2 weeks before start of protocol-specified therapy, with the exception of intrathecal chemotherapy, dexamethasone, and oral small molecule inhibitors such as BTK-inhibitor, PI3K-inhibitor, or Bcl-2-inhibitor, which are allowed until the start of protocol-specified therapy). In addition, any subject whose organ toxicity (excluding hematologic) from prior treatment has not resolved to no more than CTCAE grade 1.
8. Radiotherapy within 2 weeks before the start of protocol-specified therapy.
9. Abnormal screening laboratory values as defined as following: a) ALT (SGOT) and/or ALT (SGPT) and/or ALP > or =5 x upper limit of normal (ULN); b) Total bilirubin > or = 1.5 x ULN, unless due to Gilbert's disease; c) Creatinine > or = 2.0 x ULN or creatinine clearance <50 mL/min (calculated).
10. Known infection with human immunodeficiency virus (HIV) or chronic infection with hepatitis B virus (HBsAg positive) or hepatitis C virus (anti-HCV positive).
11. Patient is pregnant or breast feeding.
12. Woman of childbearing potential and is not willing to use 2 highly effective methods of contraception while receiving protocol-specified therapy and for an additional 24 hours after the last dose of protocol-specified therapy.
13. Male who has a female partner of childbearing potential, and is not willing to use 2 highly effective forms of contraception while receiving protocol-specified therapy and for at least an additional 24 hours after the last dose of protocol-specified therapy.
14. Male who has a pregnant partner, and is not willing to use a condom during sexual activity while receiving protocol-specified therapy and for 3 months after the last dose of protocol-specified therapy.
15. Currently receiving treatment in another investigational device or drug study.
16. Subject previously treated with blinatumomab.
17. History or evidence of any other clinically significant disorder, condition or disease (with the exception of those outlined above) that, in the opinion of the Principal Investigator would pose a risk to subject safety or interfere with the study evaluation, procedures or completion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2017-06-22 (Actual); Primary Completion 2022-02-11 (Actual); Study Completion 2022-02-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Philip A. Thompson, MBBS, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Thompson PA, Jiang X, Banerjee P, Basar R, Garg N, Chen K, Kaplan M, Nandivada V, Cortes AKN, Ferrajoli A, Keating MJ, Peterson CB, Andreeff M, Rezvani K, Wierda WG. A phase two study of high dose blinatumomab in Richter's syndrome. Leukemia. 2022 Sep;36(9):2228-2232. doi: 10.1038/s41375-022-01649-3. Epub 2022 Aug 8. PMID 35941212
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Ibrutinib, Nivolumab and Blinatumomab
Started | 9
Completed | 9
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Ibrutinib, Nivolumab and Blinatumomab
Number analyzed (Participants) | 9
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 4
  >=65 years | 5
Age, Continuous [Median (Full Range); unit: years] | 66 [50 to 76]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 7
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 9

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With a Response
Description: Response is defined as complete remission (CR) plus partial remission (PR). Complete Remission (CR) is Lymph nodes None >/= 1.5 cm, Spleen size < 13 cm; normal liver size, the absence of constitutional symptoms, normal circulating lymphocyte count, platelets >/= 100 x 10^9/L, Hemoglobin >/= 11.0 g/dL (absence of transfusion and without erythropoietin) and marrow normocellular, no CLL cells and no B-lymphoid nodules. Partial Remission (PR) is any two of the following must decrease >/= 50% from baseline: lymph nodes, Liver and/or spleen size, circulating lymphocyte count in addition to one of the following: platelets >/= 100 x 10^9/L or >/= 50% increase from baseline, Hemoglobin >/= 11.0 g/dL or >/= 50% increase from baseline or marrow presence of CLL cells, or of B-lymphoid nodules, or not done.
Time Frame: 2 months
Measure: Count of Participants; unit: Participants
Arm/Group | Ibrutinib, Nivolumab and Blinatumomab
Number analyzed (Participants) | 9
Participants | 2

2. Secondary Outcome: Number of Participants to Achieve Complete Remission
Description: Complete Remission is defined as: Complete Remission (CR) is Lymph nodes None >/= 1.5 cm, Spleen size < 13 cm; normal liver size, the absence of constitutional symptoms, normal circulating lymphocyte count, platelets >/= 100 x 10^9/L, Hemoglobin >/= 11.0 g/dL (absence of transfusion and without erythropoietin) and marrow normocellular, no CLL cells and no B-lymphoid nodules.
Time Frame: Up to 4 years, 8 months
Measure: Count of Participants; unit: Participants
Arm/Group | Ibrutinib, Nivolumab and Blinatumomab
Number analyzed (Participants) | 9
Participants | 1

3. Secondary Outcome: Progression Free Survival
Description: Time from date of treatment start until the date of first objective documentation of disease-relapse.
Time Frame: Up to 4 years, 8 months
Measure: Median (Full Range); unit: months
Arm/Group | Ibrutinib, Nivolumab and Blinatumomab
Number analyzed (Participants) | 2
months | 1.9 [1 to 17]

4. Secondary Outcome: Overall Survival
Description: Time from date of treatment start until date of death due to any cause or last Follow-up.
Time Frame: Up to 4 years, 8 Months
Measure: Median (Full Range); unit: Months
Arm/Group | Ibrutinib, Nivolumab and Blinatumomab
Number analyzed (Participants) | 9
Months | 10.3 [5 to 48]

ADVERSE EVENTS:
Time Frame: Up to 4 years, 8 months
Arm/Group | Ibrutinib, Nivolumab and Blinatumomab
All-Cause Mortality (participants affected / at risk) | 0/9
Serious Adverse Events (participants affected / at risk) | 9/9
Other Adverse Events (participants affected / at risk) | 9/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ibrutinib, Nivolumab and Blinatumomab (N=9)
Cytokine Release Syndrome (Immune system disorders) | 1 (1)
Hypercalcemia (Metabolism and nutrition disorders) | 2 (2)
Fracture (Injury, poisoning and procedural complications) | 1 (1)
Nervous System Disorder (Nervous system disorders) | 1 (1)
Creatinine Increased (Investigations) | 1 (1)
Lung Infection (Infections and infestations) | 3 (3)
Chills (General disorders) | 1 (1)
Fatigue (General disorders) | 1 (1)
Hypotension (Vascular disorders) | 1 (1)
Metabolism and nutrition disorders - Other, specify (Metabolism and nutrition disorders) | 1 (1)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Fever (General disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ibrutinib, Nivolumab and Blinatumomab (N=9)
Abdominal distension (Gastrointestinal disorders) | 1 (1)
Alanine aminotransferase increased (Investigations) | 2 (2)
Alkaline phosphatase increased (Investigations) | 3 (3)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Anorexia (Gastrointestinal disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Blood bilirubin increased (Investigations) | 1 (1)
Bruising (Skin and subcutaneous tissue disorders) | 1 (1)
Chills (General disorders) | 1 (1)
Confusion (Psychiatric disorders) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Creatinine increased (Investigations) | 2 (2)
Cytokine release syndrome (Immune system disorders) | 2 (2)
Dysgeusia (Nervous system disorders) | 1 (1)
Dysphasia (Nervous system disorders) | 1 (1)
Edema (General disorders) | 2 (3)
Erectile dysfunction (Reproductive system and breast disorders) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1)
Fatigue (General disorders) | 4 (5)
Fever (General disorders) | 5 (6)
Gastrointestinal disorders (Gastrointestinal disorders) | 1 (1)
General disorders and administration site conditions (General disorders) | 2 (3)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Hearing impaired (Ear and labyrinth disorders) | 1 (1)
Hypercalcemia (Metabolism and nutrition disorders) | 3 (3)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (1)
Hypermagnesemia (Metabolism and nutrition disorders) | 1 (1)
Hypertension (Vascular disorders) | 2 (3)
Hyperuricemia (Metabolism and nutrition disorders) | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 2 (2)
Hypocalcemia (Metabolism and nutrition disorders) | 2 (2)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 2 (3)
Hypophosphatemia (Metabolism and nutrition disorders) | 1 (1)
Hypotension (Vascular disorders) | 1 (1)
Investigations (Investigations) | 3 (12)
Lung infection (Infections and infestations) | 3 (4)
Metabolism and nutrition disorders (Metabolism and nutrition disorders) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Nervous system disorders (Nervous system disorders) | 1 (1)
Oral dysesthesia (Gastrointestinal disorders) | 1 (1)
Paresthesia (Nervous system disorders) | 1 (2)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
cough (Gastrointestinal disorders) | 1 (1)
Pain (General disorders) | 1 (1)
Respiratory, thoracic and mediastinal disorders (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 2 (2)
Skin and subcutaneous tissue disorders (Skin and subcutaneous tissue disorders) | 1 (2)
Testicular disorder (Reproductive system and breast disorders) | 1 (1)
Tremor (Nervous system disorders) | 3 (3)
Weight gain (Investigations) | 1 (1)
Weight loss (Investigations) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-03-08): https://cdn.clinicaltrials.gov/large-docs/34/NCT03121534/Prot_SAP_000.pdf